CLINICAL TRIAL: NCT00207870
Title: Comparison of Crossed Pin Versus Lateral-Entry Pin Fixation for Type II Supracondylar Fractures in Children: A Prospective, Randomized Trial
Brief Title: Type II Supracondylar Fractures in Children
Status: Withdrawn | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: Type II Supracondylar FX
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Type II Supracondylar Fractures
Keywords: Type II Supracondylar Fracture; Orthopaedics

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Supracondylar fractures are the most common elbow fractures in children. In the current orthopedic literature crossed pinning and lateral-only entry techniques are co-gold standards of operative treatment. The crossed pinning technique has been shown to be biomechanically superior especially under torsional loading but has a higher incidence of iatrogenic injury to the ulnar nerve. All studies comparing these techniques to date have been either biomechanical or retrospective in nature. A randomized, controlled, prospective study comparing these two popular techniques has not been performed.

The purpose of this study is to prospectively evaluate the amount of displacement incurred when treating type III supracondylar humerus fractures in children with crossed pinning versus lateral-entry only technique. Overall complication rate, loss of reduction, iatrogenic neurovascular injury, and pin tract infection rates between the two cohorts will be evaluated. The study population will comprise all patients less than ten years of age presenting to Scottish Rite Hospital during the study period with a type III supracondylar fracture managed by the Children's Healthcare of Atlanta Orthopedic Group. All patients will be randomized to one specific treatment arm based on surgeon preference established at the onset of the study. The hypothesis to be tested is that no difference in amount of displacement or overall complication rate is present between these two techniques. Radiographic parameters measured pre-operatively, immediately post-operatively and four weeks post-operatively will be quantitatively evaluated and compared. Chart reviews to determine complications during the treatment period will be made. Pre-study power analysis and post-study statistical analysis will be performed.

DETAILED DESCRIPTION:
Pre-operative consent forms for study participation will be reviewed with all families at the time of the pre-operative visit. Screening will be performed at the time of evaluation in the emergency room. Patients will be assigned to a particular group based on the surgeon that performs their surgery. Each surgeon at the onset of the study will commit to one technique of operative management with the understanding that this technique may be abandoned by the surgeon in any case where it is felt to be inadequate. Changing technique will be considered a failure of the technique. Data regarding the treatment will be collected from the chart and x-rays at the time of treatment and at follow up visits in the orthopedic office.

ELIGIBILITY:
Inclusion Criteria:

* Closed, Gartland's type III extension supracondylar humerus fractures requiring closed reduction and pinning.

Exclusion Criteria:

* Age greater than ten
* Open fracture
* Need for open reduction in the operating room
* Need for vascular repair of the ipsilateral extremity

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all patients less than 10 with a supracondylar fx
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Blanco, MD, Principal Investigator — Children's Orthopaedics of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia, United States